CLINICAL TRIAL: NCT01772108
Title: A Randomized Study of the MitraClip Device in Heart Failure Patients With Clinically Significant Functional Mitral Regurgitation
Acronym: RESHAPE-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As recruitment rate was lower than anticipated
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-513
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Diseases
Keywords: Heart Valve Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MitraClip Device (Experimental): Subjects randomized to the Device group will undergo the MitraClip procedure in addition to optimal standard medical therapy.
  Interventions: Device: MitraClip
- Control (No Intervention): Subjects randomized to the Control group will receive optimal standard of care therapy alone.

INTERVENTIONS:
Device: MitraClip — The MitraClip System includes a MitraClip device, a Steerable Guide Catheter, and a MitraClip Delivery System that enables placement of the MitraClip device on the mitral valve leaflets
  Arms: MitraClip Device

SUMMARY:
This trial is a randomized study of the MitraClip device in heart failure patients with clinically significant functional mitral regurgitation. A hierarchical composite of all-cause mortality and recurrent heart failure hospitalizations is hypothesized to occur at a lower rate with the use of the MitraClip device in addition to optimal standard medical therapy compared to optimal standard of care therapy alone.

DETAILED DESCRIPTION:
This study is a clinical evaluation of the safety and effectiveness of the MitraClip System in the treatment of clinically significant functional mitral regurgitation in patients with chronic heart failure. The objective was to further study the safety and effectiveness of the MitraClip System for the treatment of clinically significant functional mitral regurgitation in New York Heart Association Functional Class III or IV chronic heart failure patients.

Due to lower than expected recruitment rate, Abbott Vascular sponsorship of the trial was terminated early.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 90 years old
* Clinically significant functional mitral regurgitation (moderate-to-severe or severe mitral regurgitation), as defined by European Association of Echocardiography, within 90 days prior to randomization and confirmed by the Echocardiography Core Laboratory
* Assessed by the investigator to be on optimal standard of care therapy for heart failure for at least 4 weeks with no dose changes of heart failure drugs (with the exception of diuretics) during the last 2 weeks immediately prior to randomization
* Documented New York Heart Association Class III or Class IV heart failure, despite optimal standard of care therapy, within 90 days preceding randomization
* Minimum of one documented hospitalization (acute care admission or emergency room visit) for heart failure within 12 months preceding randomization OR values of at least 350 pg/mL for BNP or at least 1400 pg/mL for NT-proBNP after optimal medical and/or device management within 90 days preceding randomization
* Left ventricular ejection fraction (LVEF) ≥15% and ≤40% determined by transthoracic echocardiogram within 90 days prior to randomization and confirmed by the Echocardiography Core Laboratory
* Left ventricular end diastolic diameter (LVEDD) ≥55 mm determined by transthoracic echocardiogram within 90 days prior to randomization and confirmed by the Echocardiography Core Laboratory
* Patient is ambulatory and able to perform a 6MWT with the only limiting factor(s) being due to cardiovascular fitness
* Subject agrees to return for all required post-procedure follow-up visits
* The subject has been informed of the nature of the study and agrees to the study's provisions, including the possibility of randomization to the Control group, and has provided written informed consent as approved by the respective clinical site's Ethics Committee

Exclusion Criteria:

* Mitral regurgitation is primarily due to degenerative disease of the mitral valve apparatus (Degenerative mitral regurgitation), as determined by transesophageal echocardiography
* Status 1 heart transplant or prior orthotopic heart transplantation
* Introduction of a new heart failure drug class within the last 4 weeks prior to randomization
* Cardiovascular hospitalization within the last 2 weeks immediately prior to randomization
* Evidence of acute coronary syndrome, transient ischemic attack or stroke within 90 days prior to randomization
* Any percutaneous cardiovascular intervention, carotid surgery, cardiovascular surgery or atrial fibrillation ablation within 90 days prior to randomization
* Implant of any rhythm management device (i.e., pacemaker, Cardiac Resynchronization Therapy with or without cardioverter-defibrillator (CRT or CRT-D), or Implantable Cardioverter Defibrillator (ICD) within 90 days prior to randomization, or revision of any implanted rhythm management device within 90 days prior to randomization
* Need for any cardiovascular surgery
* Mitral valve surgery is considered a therapeutic option for the subject
* Renal replacement therapy
* Uncontrolled hypertension (i.e., BP >180 mmHg systolic and/or >105 mmHg diastolic) or hypotension (i.e., BP <90 mmHg systolic)
* Unstable angina pectoris as judged by the investigator, other clinically significant uncorrected valvular disease or left ventricular outflow obstruction, obstructive cardiomyopathy, poorly controlled fast atrial fibrillation or flutter, poorly controlled symptomatic brady- or tachyarrhythmias
* 6MWT distance >450 meters
* Mitral Valve Area (MVA) by planimetry <4.0 cm2; if MVA by planimetry is not measurable, pressure half-time measurement is acceptable; MVA must be confirmed by the Echocardiography Core Laboratory
* Leaflet anatomy which may preclude MitraClip device implantation, proper device positioning on the leaflets, or sufficient reduction in mitral regurgitation that may include:

  * Evidence of calcification in the grasping area
  * Presence of significant cleft in the grasping area
  * Lack of both primary and secondary chordal support in the grasping area
  * Prior mitral valve surgery
  * Coaptation length ≤2 mm
  * Leaflet mobility length <1 cm
* Presence of an IVC filter in the femoral vein that would interfere with the delivery catheter, or ipsilateral deep vein thrombosis (DVT) is present
* Contraindication to transseptal catheterization
* Subjects in whom transesophageal echocardiography is contraindicated
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (i.e., noncompliant, perforated)
* Presence of any of the following:

  * Severe aortic stenosis (aortic valve area <1.0 cm2) or severe aortic regurgitation
  * Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis)
  * Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
  * Hemodynamic instability requiring inotropic support or mechanical heart circulatory support
* Active infections requiring current antibiotic therapy
* Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically
* Severe right ventricular failure or severe tricuspid regurgitation
* History of bleeding diathesis or coagulopathy or subject who refuses blood transfusions
* Pregnant or planning pregnancy within next 12 months. Note: Female patients of childbearing potential need to have a negative pregnancy test performed within 14 days prior to randomization and be adherent to an accepted method of contraception
* Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the investigator
* Currently participating in another therapeutic or interventional heart failure trial, or in any trial of an unapproved drug or device (Subjects participating in observational studies or registries may be considered as eligible)
* Subject belongs to a vulnerable population per investigator's judgment or subject has any kind of disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Hierarchical composite of all-cause mortality and recurrent heart failure hospitalizations | two years
  The analysis will be carried out when the last patient completes 12-month follow-up. All follow-up, up to 24 months, will be included in the analysis.

SECONDARY OUTCOMES:
Composite of all-cause mortality, stroke, myocardial infarction, new need for renal replacement therapy, and non-elective cardiovascular surgery for device related complications in the Device group at 30 days | 30 days
Mitral regurgitation severity reduction to mild or mild-to-moderate at 12 months | 12 months
Change in Left Ventricular End Diastolic Volume (LVEDV) at 12 months over baseline | 12 months
Change in Left Ventricular End Systolic Volume (LVESV) at 12 months over baseline | 12 months
Change in 6 Minute Walk Test (6MWT) distance at 12 months over baseline | 12 months
Change in Quality of Life (QoL) score, as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ), at 12 months over baseline | 12 months
New York Heart Association (NYHA) Functional Class I/II at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ponikowski, MD, PhD, Principal Investigator — Military Hospital, Medical University, Wroclaw, Poland
Locations (29):
- Allgemein öffentliches Krankenhaus Elisabethinen Linz, Linz, Fadingerstraße 1, Austria
- UZA, Edegem, Belgium
- Denmark (3):
  - Skejby Sykehus/Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense
- Helsinki University Hospital, Helsinki, Finland
- Germany (10):
  - Universitätsklinikum der RWTH - Aachen, Aachen
  - Herz-Zentrum, Bad Krozingen
  - Charité - Universitätsmedizin Berlin, Berlin
  - Evangelish-Freikirchliches Krankenhaus, Bernau, Bernau
  - Herzzentrum Göttingen Universitätsmedizin, Göttingen, Göttingen
  - Asklepios Klinik St Georg, Hamburg, Hamburg
  - Kardiologische Gemeinschaftspraxis Mathey-Schofer, Hamburg, Hamburg
  - Universitäre Herzzentrum, Hamburg, Hamburg
  - Uni-Klinikum Heidelberg, Heidelberg
  - Johannes Gütenberg University, Mainz, Mainz
- Italy (5):
  - Spedali Civili di Brescia, Brescia
  - Ospedale Ferrarotto Alessi, Catania, Catania
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Raffaele, Milano, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St Antonius Ziekenhuis, Nieuwegein, Nieuwegein
- Hospital Sant Creu y Sant Pau,, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Stockholm, Sweden
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Universitäts Spital Zürich, Zurich

REFERENCES:
- [Background] McGee EC Jr. Should moderate or greater mitral regurgitation be repaired in all patients with LVEF <30%? Surgery, mitral regurgitation, and heart failure: the valves are all repairable but the patients are not. Circ Heart Fail. 2008 Nov;1(4):285-9. doi: 10.1161/CIRCHEARTFAILURE.108.800185. No abstract available. PMID 19808304
- [Background] Fruhwald F, Pieske B. Left ventricular remodelling in systolic heart failure using ivabradine. Slower is smaller is better? Eur Heart J. 2011 Oct;32(20):2481-2. doi: 10.1093/eurheartj/ehr317. Epub 2011 Aug 29. No abstract available. PMID 21875857
- [Background] Zannad F. Acute heart failure syndromes: the 'Cinderella' of heart failure research. European Journal Supplements. 2005 April 7;(suppl B):B8-B127.
- [Background] Martinez-Selles M, Garcia Robles JA, Prieto L, Serrano JA, Munoz R, Frades E, Almendral J. Annual rates of admission and seasonal variations in hospitalizations for heart failure. Eur J Heart Fail. 2002 Dec;4(6):779-86. doi: 10.1016/s1388-9842(02)00116-2. PMID 12453550
- [Background] Reducing Heart Failure Hospitalization. Genesis Heart Institute. http://www.genesishealth.com/ghi/news/hf_hospitalization 2011 Oct 18.
- [Background] Pino PG, Galati A, Terranova A. Functional mitral regurgitation in heart failure. J Cardiovasc Med (Hagerstown). 2006 Jul;7(7):514-23. doi: 10.2459/01.JCM.0000234770.88701.75. PMID 16801813
- [Background] American Heart Association/American College of Cardiology (AHA/ACC) 2009 update HF guidelines.
- [Background] Linde C, Mealing S, Hawkins N, Eaton J, Brown B, Daubert JC; REVERSE study group. Cost-effectiveness of cardiac resynchronization therapy in patients with asymptomatic to mild heart failure: insights from the European cohort of the REVERSE (Resynchronization Reverses remodeling in Systolic Left Ventricular Dysfunction). Eur Heart J. 2011 Jul;32(13):1631-9. doi: 10.1093/eurheartj/ehq408. Epub 2010 Nov 25. PMID 21112898
- [Background] Lebrun F, Lancellotti P, Pierard LA. Quantitation of functional mitral regurgitation during bicycle exercise in patients with heart failure. J Am Coll Cardiol. 2001 Nov 15;38(6):1685-92. doi: 10.1016/s0735-1097(01)01605-9. PMID 11704381
- [Background] Schmitto JD, Lee LS, Mokashi SA, Bolman RM 3rd, Cohn LH, Chen FY. Functional mitral regurgitation. Cardiol Rev. 2010 Nov-Dec;18(6):285-91. doi: 10.1097/CRD.0b013e3181e8e648. PMID 20926937
- [Background] Michelena HI, Bichara VM, Margaryan E, Forde I, Topilsky Y, Suri R, Enriquez-Sarano M. Progress in the treatment of severe mitral regurgitation. Rev Esp Cardiol. 2010 Jul;63(7):820-31. doi: 10.1016/s1885-5857(10)70167-5. English, Spanish. PMID 20609316
- [Background] Southard J, and Rogers J. Current Catheter-Based Treatments of Functional Mitral Regurgitation. Cardiac Interventions. 2007 June.
- [Background] Delling FN, Kang LL, Yeon SB, Kissinger KV, Goddu B, Manning WJ, Han Y. CMR predictors of mitral regurgitation in mitral valve prolapse. JACC Cardiovasc Imaging. 2010 Oct;3(10):1037-45. doi: 10.1016/j.jcmg.2010.06.016. PMID 20947049
- [Background] Otsuji Y, Handschumacher MD, Schwammenthal E, Jiang L, Song JK, Guerrero JL, Vlahakes GJ, Levine RA. Insights from three-dimensional echocardiography into the mechanism of functional mitral regurgitation: direct in vivo demonstration of altered leaflet tethering geometry. Circulation. 1997 Sep 16;96(6):1999-2008. doi: 10.1161/01.cir.96.6.1999. PMID 9323092
- [Background] Carabello BA, Nakano K, Corin W, Biederman R, Spann JF Jr. Left ventricular function in experimental volume overload hypertrophy. Am J Physiol. 1989 Apr;256(4 Pt 2):H974-81. doi: 10.1152/ajpheart.1989.256.4.H974. PMID 2523200
- [Background] Digitalis Investigation Group. The effect of digoxin on mortality and morbidity in patients with heart failure. N Engl J Med. 1997 Feb 20;336(8):525-33. doi: 10.1056/NEJM199702203360801. PMID 9036306
- [Background] Taylor AL, Ziesche S, Yancy C, Carson P, D'Agostino R Jr, Ferdinand K, Taylor M, Adams K, Sabolinski M, Worcel M, Cohn JN; African-American Heart Failure Trial Investigators. Combination of isosorbide dinitrate and hydralazine in blacks with heart failure. N Engl J Med. 2004 Nov 11;351(20):2049-57. doi: 10.1056/NEJMoa042934. Epub 2004 Nov 8. PMID 15533851
- [Background] Breithardt OA, Sinha AM, Schwammenthal E, Bidaoui N, Markus KU, Franke A, Stellbrink C. Acute effects of cardiac resynchronization therapy on functional mitral regurgitation in advanced systolic heart failure. J Am Coll Cardiol. 2003 Mar 5;41(5):765-70. doi: 10.1016/s0735-1097(02)02937-6. PMID 12628720
- [Background] Kanzaki H, Bazaz R, Schwartzman D, Dohi K, Sade LE, Gorcsan J 3rd. A mechanism for immediate reduction in mitral regurgitation after cardiac resynchronization therapy: insights from mechanical activation strain mapping. J Am Coll Cardiol. 2004 Oct 19;44(8):1619-25. doi: 10.1016/j.jacc.2004.07.036. PMID 15489094
- [Background] Abraham WT. Cardiac resynchronization therapy. Prog Cardiovasc Dis. 2006 Jan-Feb;48(4):232-8. doi: 10.1016/j.pcad.2005.11.001. PMID 16517245
- [Background] Auricchio A, Abraham WT. Cardiac resynchronization therapy: current state of the art: cost versus benefit. Circulation. 2004 Jan 27;109(3):300-7. doi: 10.1161/01.CIR.0000115583.20268.E1. No abstract available. PMID 14744954
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W; MADIT-CRT Trial Investigators. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009 Oct 1;361(14):1329-38. doi: 10.1056/NEJMoa0906431. Epub 2009 Sep 1. PMID 19723701
- [Background] Linde C, Abraham WT, Gold MR, St John Sutton M, Ghio S, Daubert C; REVERSE (REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction) Study Group. Randomized trial of cardiac resynchronization in mildly symptomatic heart failure patients and in asymptomatic patients with left ventricular dysfunction and previous heart failure symptoms. J Am Coll Cardiol. 2008 Dec 2;52(23):1834-1843. doi: 10.1016/j.jacc.2008.08.027. Epub 2008 Nov 7. PMID 19038680
- [Background] McAlister FA, Ezekowitz J, Hooton N, Vandermeer B, Spooner C, Dryden DM, Page RL, Hlatky MA, Rowe BH. Cardiac resynchronization therapy for patients with left ventricular systolic dysfunction: a systematic review. JAMA. 2007 Jun 13;297(22):2502-14. doi: 10.1001/jama.297.22.2502. PMID 17565085
- [Background] Heart Failure Society of America; Lindenfeld J, Albert NM, Boehmer JP, Collins SP, Ezekowitz JA, Givertz MM, Katz SD, Klapholz M, Moser DK, Rogers JG, Starling RC, Stevenson WG, Tang WH, Teerlink JR, Walsh MN. HFSA 2010 Comprehensive Heart Failure Practice Guideline. J Card Fail. 2010 Jun;16(6):e1-194. doi: 10.1016/j.cardfail.2010.04.004. PMID 20610207
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur Heart J. 2008 Oct;29(19):2388-442. doi: 10.1093/eurheartj/ehn309. Epub 2008 Sep 17. No abstract available. PMID 18799522
- [Background] Haddad H, Isaac D, Legare JF, Pflugfelder P, Hendry P, Chan M, Cantin B, Giannetti N, Zieroth S, White M, Warnica W, Doucette K, Rao V, Dipchand A, Cantarovich M, Kostuk W, Cecere R, Charbonneau E, Ross H, Poirier N. Canadian Cardiovascular Society Consensus Conference update on cardiac transplantation 2008: Executive Summary. Can J Cardiol. 2009 Apr;25(4):197-205. doi: 10.1016/s0828-282x(09)70061-3. No abstract available. PMID 19340342
- [Background] Mehra MR, Kobashigawa J, Starling R, Russell S, Uber PA, Parameshwar J, Mohacsi P, Augustine S, Aaronson K, Barr M. Listing criteria for heart transplantation: International Society for Heart and Lung Transplantation guidelines for the care of cardiac transplant candidates--2006. J Heart Lung Transplant. 2006 Sep;25(9):1024-42. doi: 10.1016/j.healun.2006.06.008. No abstract available. PMID 16962464
- [Background] Arnold JM, Liu P, Demers C, Dorian P, Giannetti N, Haddad H, Heckman GA, Howlett JG, Ignaszewski A, Johnstone DE, Jong P, McKelvie RS, Moe GW, Parker JD, Rao V, Ross HJ, Sequeira EJ, Svendsen AM, Teo K, Tsuyuki RT, White M; Canadian Cardiovascular Society. Canadian Cardiovascular Society consensus conference recommendations on heart failure 2006: diagnosis and management. Can J Cardiol. 2006 Jan;22(1):23-45. doi: 10.1016/s0828-282x(06)70237-9. PMID 16450016
- [Background] Hunt SA; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure). ACC/AHA 2005 guideline update for the diagnosis and management of chronic heart failure in the adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure). J Am Coll Cardiol. 2005 Sep 20;46(6):e1-82. doi: 10.1016/j.jacc.2005.08.022. No abstract available. PMID 16168273
- [Background] De Bonis M, Taramasso M, Verzini A, Ferrara D, Lapenna E, Calabrese MC, Grimaldi A, Alfieri O. Long-term results of mitral repair for functional mitral regurgitation in idiopathic dilated cardiomyopathy. Eur J Cardiothorac Surg. 2012 Oct;42(4):640-6. doi: 10.1093/ejcts/ezs078. Epub 2012 Mar 23. PMID 22447810
- [Background] Grossi EA, Crooke GA, DiGiorgi PL, Schwartz CF, Jorde U, Applebaum RM, Ribakove GH, Galloway AC, Grau JB, Colvin SB. Impact of moderate functional mitral insufficiency in patients undergoing surgical revascularization. Circulation. 2006 Jul 4;114(1 Suppl):I573-6. doi: 10.1161/CIRCULATIONAHA.105.001230. PMID 16820640
- [Background] Thourani VH, Weintraub WS, Guyton RA, Jones EL, Williams WH, Elkabbani S, Craver JM. Outcomes and long-term survival for patients undergoing mitral valve repair versus replacement: effect of age and concomitant coronary artery bypass grafting. Circulation. 2003 Jul 22;108(3):298-304. doi: 10.1161/01.CIR.0000079169.15862.13. Epub 2003 Jun 30. PMID 12835220
- [Background] Bouchard D, Pellerin M, Carrier M, Perrault LP, Page P, Hebert Y, Cartier R, Dyrda I, Pelletier LC. Results following valve replacement for ischemic mitral regurgitation. Can J Cardiol. 2001 Apr;17(4):427-31. PMID 11329543
- [Background] Wu AH, Aaronson KD, Bolling SF, Pagani FD, Welch K, Koelling TM. Impact of mitral valve annuloplasty on mortality risk in patients with mitral regurgitation and left ventricular systolic dysfunction. J Am Coll Cardiol. 2005 Feb 1;45(3):381-7. doi: 10.1016/j.jacc.2004.09.073. PMID 15680716
- [Background] Levine RA, Schwammenthal E. Ischemic mitral regurgitation on the threshold of a solution: from paradoxes to unifying concepts. Circulation. 2005 Aug 2;112(5):745-58. doi: 10.1161/CIRCULATIONAHA.104.486720. No abstract available. PMID 16061756
- [Background] Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2008 focused update incorporated into the ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to revise the 1998 guidelines for the management of patients with valvular heart disease). Endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2008 Sep 23;52(13):e1-142. doi: 10.1016/j.jacc.2008.05.007. No abstract available. PMID 18848134
- [Background] A Class IIb; Level of Evidence C recommendation is defined as: "Recommendation's usefulness/efficacy less well established. Only diverging expert opinion, case studies, or standard of care."
- [Background] Feldman T, Foster E, Glower DD, Kar S, Rinaldi MJ, Fail PS, Smalling RW, Siegel R, Rose GA, Engeron E, Loghin C, Trento A, Skipper ER, Fudge T, Letsou GV, Massaro JM, Mauri L; EVEREST II Investigators. Percutaneous repair or surgery for mitral regurgitation. N Engl J Med. 2011 Apr 14;364(15):1395-406. doi: 10.1056/NEJMoa1009355. Epub 2011 Apr 4. PMID 21463154
- [Background] Auricchio A, Schillinger W, Meyer S, Maisano F, Hoffmann R, Ussia GP, Pedrazzini GB, van der Heyden J, Fratini S, Klersy C, Komtebedde J, Franzen O; PERMIT-CARE Investigators. Correction of mitral regurgitation in nonresponders to cardiac resynchronization therapy by MitraClip improves symptoms and promotes reverse remodeling. J Am Coll Cardiol. 2011 Nov 15;58(21):2183-9. doi: 10.1016/j.jacc.2011.06.061. PMID 22078424
- [Background] Lancellotti P, Moura L, Pierard LA, Agricola E, Popescu BA, Tribouilloy C, Hagendorff A, Monin JL, Badano L, Zamorano JL; European Association of Echocardiography. European Association of Echocardiography recommendations for the assessment of valvular regurgitation. Part 2: mitral and tricuspid regurgitation (native valve disease). Eur J Echocardiogr. 2010 May;11(4):307-32. doi: 10.1093/ejechocard/jeq031. PMID 20435783
- [Background] Optimal medical and/or device therapy includes optimal stabilization of symptoms with the use of appropriate evidence-based therapies including medicines, revascularization, and cardiac resynchronization therapy with or without cardioverter-defibrillator as indicated, per the European Society of Cardiology (ESC) guidelines
- [Background] Enriquez-Sarano M, Loulmet DF, Burkhoff D. The conundrum of functional mitral regurgitation in chronic heart failure. J Am Coll Cardiol. 2008 Jan 29;51(4):487-9. doi: 10.1016/j.jacc.2007.09.046. No abstract available. PMID 18222361
- [Background] Felker GM, Pang PS, Adams KF, Cleland JG, Cotter G, Dickstein K, Filippatos GS, Fonarow GC, Greenberg BH, Hernandez AF, Khan S, Komajda M, Konstam MA, Liu PP, Maggioni AP, Massie BM, McMurray JJ, Mehra M, Metra M, O'Connell J, O'Connor CM, Pina IL, Ponikowski P, Sabbah HN, Teerlink JR, Udelson JE, Yancy CW, Zannad F, Gheorghiade M; International AHFS Working Group. Clinical trials of pharmacological therapies in acute heart failure syndromes: lessons learned and directions forward. Circ Heart Fail. 2010 Mar;3(2):314-25. doi: 10.1161/CIRCHEARTFAILURE.109.893222. No abstract available. PMID 20233993
- [Background] Pitt B, Poole-Wilson PA, Segal R, Martinez FA, Dickstein K, Camm AJ, Konstam MA, Riegger G, Klinger GH, Neaton J, Sharma D, Thiyagarajan B. Effect of losartan compared with captopril on mortality in patients with symptomatic heart failure: randomised trial--the Losartan Heart Failure Survival Study ELITE II. Lancet. 2000 May 6;355(9215):1582-7. doi: 10.1016/s0140-6736(00)02213-3. PMID 10821361
- [Background] Cohn JN, Tognoni G; Valsartan Heart Failure Trial Investigators. A randomized trial of the angiotensin-receptor blocker valsartan in chronic heart failure. N Engl J Med. 2001 Dec 6;345(23):1667-75. doi: 10.1056/NEJMoa010713. PMID 11759645
- [Background] Pfeffer MA, Swedberg K, Granger CB, Held P, McMurray JJ, Michelson EL, Olofsson B, Ostergren J, Yusuf S, Pocock S; CHARM Investigators and Committees. Effects of candesartan on mortality and morbidity in patients with chronic heart failure: the CHARM-Overall programme. Lancet. 2003 Sep 6;362(9386):759-66. doi: 10.1016/s0140-6736(03)14282-1. PMID 13678868
- [Background] Effect of metoprolol CR/XL in chronic heart failure: Metoprolol CR/XL Randomised Intervention Trial in Congestive Heart Failure (MERIT-HF). Lancet. 1999 Jun 12;353(9169):2001-7. PMID 10376614
- [Background] Kindermann M, Hennen B, Jung J, Geisel J, Bohm M, Frohlig G. Biventricular versus conventional right ventricular stimulation for patients with standard pacing indication and left ventricular dysfunction: the Homburg Biventricular Pacing Evaluation (HOBIPACE). J Am Coll Cardiol. 2006 May 16;47(10):1927-37. doi: 10.1016/j.jacc.2005.12.056. Epub 2006 Apr 24. PMID 16697307
- [Background] Nishimura RA, Schaff HV: Mitral regurgitation: timing of surgery. In: Otto CM, Bonow RO, ed. Valvular Heart Disease: A Companion to Braunwald's Heart Disease, Philadelphia: Saunders/Elsevier; 2009:274-290.
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] The Society of Thoracic Surgeons (2005-2012). Online STS Risk Calculator: http://riskcalc.sts.org/STSWebRiskCalc273/
- [Background] Nishimura RA, Carabello BA, Faxon DP, Freed MD, Lytle BW, O'Gara PT, O'Rourke RA, Shah PM, Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS, Smith SC Jr, Jacobs AK, Buller CE, Creager MA, Ettinger SM, Krumholz HM, Kushner FG, Lytle BW, Nishimura RA, Page RL, Tarkington LG, Yancy CW Jr; American College of Cardiology/American Heart Association Task Force. ACC/AHA 2008 guideline update on valvular heart disease: focused update on infective endocarditis: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines: endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Circulation. 2008 Aug 19;118(8):887-96. doi: 10.1161/CIRCULATIONAHA.108.190377. Epub 2008 Jul 28. No abstract available. PMID 18663090
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Background] Thompson SG, Barber JA. How should cost data in pragmatic randomised trials be analysed? BMJ. 2000 Apr 29;320(7243):1197-200. doi: 10.1136/bmj.320.7243.1197. No abstract available. PMID 10784550
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Fenwick E, Claxton K, Sculpher M. Representing uncertainty: the role of cost-effectiveness acceptability curves. Health Econ. 2001 Dec;10(8):779-87. doi: 10.1002/hec.635. PMID 11747057
- [Background] National Institute for Health and Clinical Excellence (NICE) Methods for Technology Appraisal. London. 2008. http://www.nice.org.uk/media/4A6/0F/SelectedFurtherReading210708.pdf
- [Background] Leon MB, Piazza N, Nikolsky E, Blackstone EH, Cutlip DE, Kappetein AP, Krucoff MW, Mack M, Mehran R, Miller C, Morel MA, Petersen J, Popma JJ, Takkenberg JJ, Vahanian A, van Es GA, Vranckx P, Webb JG, Windecker S, Serruys PW. Standardized endpoint definitions for transcatheter aortic valve implantation clinical trials: a consensus report from the Valve Academic Research Consortium. Eur Heart J. 2011 Jan;32(2):205-17. doi: 10.1093/eurheartj/ehq406. Epub 2011 Jan 6. PMID 21216739
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Solomon SD, Dobson J, Pocock S, Skali H, McMurray JJ, Granger CB, Yusuf S, Swedberg K, Young JB, Michelson EL, Pfeffer MA; Candesartan in Heart failure: Assessment of Reduction in Mortality and morbidity (CHARM) Investigators. Influence of nonfatal hospitalization for heart failure on subsequent mortality in patients with chronic heart failure. Circulation. 2007 Sep 25;116(13):1482-7. doi: 10.1161/CIRCULATIONAHA.107.696906. Epub 2007 Aug 27. PMID 17724259
- [Background] EuroSCORE Calculator: http://www.euroscore.org/calc.html
- [Background] Pfister R, Diedrichs H, Schiedermair A, Rosenkranz S, Hellmich M, Erdmann E, Schneider CA. Prognostic impact of NT-proBNP and renal function in comparison to contemporary multi-marker risk scores in heart failure patients. Eur J Heart Fail. 2008 Mar;10(3):315-20. doi: 10.1016/j.ejheart.2008.01.009. Epub 2008 Mar 4. PMID 18304872
- [Background] Berger R, Shankar A, Fruhwald F, Fahrleitner-Pammer A, Freemantle N, Tavazzi L, Cleland JG, Pacher R. Relationships between cardiac resynchronization therapy and N-terminal pro-brain natriuretic peptide in patients with heart failure and markers of cardiac dyssynchrony: an analysis from the Cardiac Resynchronization in Heart Failure (CARE-HF) study. Eur Heart J. 2009 Sep;30(17):2109-16. doi: 10.1093/eurheartj/ehp210. Epub 2009 Jun 2. PMID 19493864
- [Background] Olsson LG, Swedberg K, Cleland JG, Spark PA, Komajda M, Metra M, Torp-Pedersen C, Remme WJ, Scherhag A, Poole-Wilson P; COMET Investigators. Prognostic importance of plasma NT-pro BNP in chronic heart failure in patients treated with a beta-blocker: results from the Carvedilol Or Metoprolol European Trial (COMET) trial. Eur J Heart Fail. 2007 Aug;9(8):795-801. doi: 10.1016/j.ejheart.2007.07.010. PMID 17693380
- [Background] Pocock SJ, Wang D, Pfeffer MA, Yusuf S, McMurray JJ, Swedberg KB, Ostergren J, Michelson EL, Pieper KS, Granger CB. Predictors of mortality and morbidity in patients with chronic heart failure. Eur Heart J. 2006 Jan;27(1):65-75. doi: 10.1093/eurheartj/ehi555. Epub 2005 Oct 11. PMID 16219658
- [Background] http://www.euroscore.org/calcold.html
- [Background] Finkelstein DM, Schoenfeld DA. Combining mortality and longitudinal measures in clinical trials. Stat Med. 1999 Jun 15;18(11):1341-54. doi: 10.1002/(sici)1097-0258(19990615)18:113.0.co;2-7. PMID 10399200
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Schillinger W, Athanasiou T, Weicken N, Berg L, Tichelbacker T, Puls M, Hunlich M, Wachter R, Helms HJ, Seipelt R, Schondube FA, Hasenfuss G. Impact of the learning curve on outcomes after percutaneous mitral valve repair with MitraClip and lessons learned after the first 75 consecutive patients. Eur J Heart Fail. 2011 Dec;13(12):1331-9. doi: 10.1093/eurjhf/hfr141. Epub 2011 Oct 24. PMID 22024027